CLINICAL TRIAL: NCT01105767
Title: Evaluating Strategies to Prevent Methicillin-resistant Staphylococcus Aureus Skin and Soft Tissue Infections in Military Trainees
Brief Title: Methicillin-resistant Staphylococcus Aureus (MRSA) Skin and Soft Tissue Infection (SSTI) Prevention in Military Trainees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: IDCRP-055
Record Dates: First submitted 2010-04-14; First posted 2010-04-16 (Estimated); Results first posted 2014-11-04 (Estimated); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Staphylococcus Aureus; MRSA Skin Infections; Staphylococcal Skin Infections
Keywords: Staphylococcus aureus; MRSA Skin Infection; Staphylococcal Skin Infections; Chlorhexidine gluconate
MeSH Terms: conditions — Staphylococcal Infections; Staphylococcal Skin Infections | interventions — chlorhexidine gluconate; Educational Status; Hygiene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 Standard (No Intervention): Trainees received a preventive medicine briefing augmented with SSTI and MRSA SSTI prevention information and personal hygiene instructions. Trainees seeking medical care for an SSTI received standardized SSTI care (e.g., antimicrobial therapy, wound management, patient education) at the Troop Medical Clinic. High-touch common surfaces within the battalion areas were cleaned with standard Environmental Protection Agency-registered disinfectants.
- Group 2 Enhanced Standard (Active Comparator): Trainees received the components of the Standard group as well as supplemental training, education and hygiene. They were instructed to take an additional 10-minute shower with soap and a wash cloth every week. They were also issued a first aid kit. Supplemental SSTI education for trainees and drill sergeants was also provided (e.g., pocket cards, posters). Drill sergeants received briefings on SSTI and skin inspection/minor wound care.
  Interventions: Other: Supplemental training, education and hygiene
- Group 3 Chlorhexidine (Active Comparator): Trainees received the components of the Standard and Enhanced Standard groups and were offered chlorhexidine body wash (4% chlorhexidine gluconate, Hibiclens®, Mӧlnlycke Heath Care, Norcross, Georgia) to use with a wash cloth after using their personal soap for the additional once-weekly shower. Trainees were provided with verbal and written/graphic instructions for use.
  Interventions: Drug: Chlorhexidine gluconate; Other: Supplemental training, education and hygiene

INTERVENTIONS:
Drug: Chlorhexidine gluconate — Self applied chlorhexidine body wash (4% chlorhexidine gluconate, Hibiclens®, Mӧlnlycke Heath Care, Norcross, Georgia) once a week to wash/cover the body (except the face and genitalia).
  Arms: Group 3 Chlorhexidine
Other: Supplemental training, education and hygiene — Supplemental SSTI education for trainees and drill sergeants included pocket cards and posters. Drill sergeants received briefings on SSTI and skin inspection/minor wound care. Trainees were instructed to take an additional 10-minute shower with soap and a wash cloth every week. They were also issued a first aid kit.
  Arms: Group 2 Enhanced Standard; Group 3 Chlorhexidine

SUMMARY:
This cluster-randomized prospective study will evaluate the effect of hygiene-based intervention strategies on the incidence of overall SSTI and MRSA-associated SSTI among military trainees. The proposed interventions used singly or in combination include standardized training and education, and weekly chlorhexidine showers.

DETAILED DESCRIPTION:
MRSA SSTIs have become endemic in congregate community settings where there is frequent close person-to-person contact, such as athletic teams, correctional facilities, and military training facilities. These infections interfere with the mission of training soldiers as they impair soldiers' ability to participate in required activities and successfully complete a training program. Hygiene-based prevention programs (e.g., hand washing, environmental disinfection, and community-based education) appear to be effective in stemming outbreaks of MRSA SSTIs and need to by systematical evaluated.

This cluster-randomized prospective study will evaluate the effect of hygiene-based intervention strategies on the incidence of overall SSTI and MRSA-associated SSTI among military trainees. The study population will be drawn from six training battalions, each consisting of an average of six companies. Each company is composed of four platoons consisting of approximately 50 trainees. Training battalions are the unit of randomization in this study and sub-clusters (platoons within companies) within each battalion will receive the same hygiene-based intervention assigned to that battalion at study start. During the proposed 20-month evaluation period, five cycles of platoons (approximately 14 weeks per cycle) will enter and exit training activities. In total, the study population will be comprised of approximately 36,000 trainees observed over a 20-month period. Each of the six battalions will receive an in-processing preventive medicine briefing augmented with MRSA prevention information based on U.S. Army Center for Health Promotion and Preventive Medicine (USACHPPM) and Centers for Disease Control and Prevention (CDC) recommendations. Additionally, trainees who seek medical care for a SSTI will receive standardized care at a SSTI clinic applying uniform practice guidance. Four of the battalions will also receive supplemental SSTI education for trainees and drill sergeants, including standardized guidance on SSTI surveillance (e.g., skin inspection) for drill sergeants; trainees will be instructed to take a 10 minute shower with soap every Sunday while in garrison; and will be issued a personal first aid kit. Two of these four battalions will be offered chlorhexidine antiseptic body wash to use during the Sunday shower. Endpoints of the evaluation (i.e., incident SSTIs among military trainees) will be captured through clinical record review at the completion of training.

ELIGIBILITY:
Inclusion Criteria:

* Trainees assigned to one of the six selected training battalions
* Trainees who present with an SSTI at the clinic or the hospital
* Provide informed consent

Exclusion Criteria:

* Fails to meet inclusion criteria

Ages: 18 Years to 42 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30209 (Actual)
Dates: Start 2010-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ellis, MD, Principal Investigator — Uniformed Services University of the Health Sciences
Locations (1):
- Usa Meddac Mach, Columbus, Georgia, United States

REFERENCES:
- [Derived] Jefferson T, Dooley L, Ferroni E, Al-Ansary LA, van Driel ML, Bawazeer GA, Jones MA, Hoffmann TC, Clark J, Beller EM, Glasziou PP, Conly JM. Physical interventions to interrupt or reduce the spread of respiratory viruses. Cochrane Database Syst Rev. 2023 Jan 30;1(1):CD006207. doi: 10.1002/14651858.CD006207.pub6. PMID 36715243
- [Derived] Jefferson T, Del Mar CB, Dooley L, Ferroni E, Al-Ansary LA, Bawazeer GA, van Driel ML, Jones MA, Thorning S, Beller EM, Clark J, Hoffmann TC, Glasziou PP, Conly JM. Physical interventions to interrupt or reduce the spread of respiratory viruses. Cochrane Database Syst Rev. 2020 Nov 20;11(11):CD006207. doi: 10.1002/14651858.CD006207.pub5. PMID 33215698
- [Derived] Johnson RC, Ellis MW, Schlett CD, Millar EV, LaBreck PT, Mor D, Elassal EM, Lanier JB, Redden CL, Cui T, Teneza-Mora N, Bishop DK, Hall ER, Bishop-Lilly KA, Merrell DS. Bacterial Etiology and Risk Factors Associated with Cellulitis and Purulent Skin Abscesses in Military Trainees. PLoS One. 2016 Oct 25;11(10):e0165491. doi: 10.1371/journal.pone.0165491. eCollection 2016. PMID 27780238
- [Derived] Millar EV, Schlett CD, Law NN, Chen WJ, D'Onofrio MJ, Bennett JW, Tribble DR, Ellis MW. Reduction in Acute Respiratory Infection Among Military Trainees: Secondary Effects of a Hygiene-Based Cluster-Randomized Trial for Skin and Soft-Tissue Infection Prevention. Infect Control Hosp Epidemiol. 2016 Sep;37(9):1118-20. doi: 10.1017/ice.2016.154. Epub 2016 Jul 8. No abstract available. PMID 27387422
- [Derived] D'Onofrio MJ, Schlett CD, Millar EV, Cui T, Lanier JB, Law NN, Tribble DR, Ellis MW. Reduction in acute gastroenteritis among military trainees: secondary effects of a hygiene-based cluster-randomized trial for skin and soft tissue infection prevention. Infect Control Hosp Epidemiol. 2015 Mar;36(3):358-60. doi: 10.1017/ice.2014.65. PMID 25695181
- [Derived] Millar EV, Chen WJ, Schlett CD, Cui T, Crawford KB, Lanier JB, Tribble DR, Ellis MW. Frequent use of chlorhexidine-based body wash associated with a reduction in methicillin-resistant Staphylococcus aureus nasal colonization among military trainees. Antimicrob Agents Chemother. 2015 Feb;59(2):943-9. doi: 10.1128/AAC.03993-14. Epub 2014 Nov 24. PMID 25421482
- [Derived] Ellis MW, Schlett CD, Millar EV, Crawford KB, Cui T, Lanier JB, Tribble DR. Prevalence of nasal colonization and strain concordance in patients with community-associated Staphylococcus aureus skin and soft-tissue infections. Infect Control Hosp Epidemiol. 2014 Oct;35(10):1251-6. doi: 10.1086/678060. Epub 2014 Aug 19. PMID 25203178
- [Derived] Ellis MW, Schlett CD, Millar EV, Wilkins KJ, Crawford KB, Morrison-Rodriguez SM, Pacha LA, Gorwitz RJ, Lanier JB, Tribble DR. Hygiene strategies to prevent methicillin-resistant Staphylococcus aureus skin and soft tissue infections: a cluster-randomized controlled trial among high-risk military trainees. Clin Infect Dis. 2014 Jun;58(11):1540-8. doi: 10.1093/cid/ciu166. Epub 2014 Mar 14. PMID 24633684

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 Standard: Trainees received a preventive medicine briefing augmented with SSTI and MRSA SSTI prevention information and personal hygiene instructions. Trainees seeking medical care for an SSTI received standardized SSTI care (e.g., antimicrobial therapy, wound management, patient education) at the Troop Medical Clinic. High-touch common surfaces within the battalion areas were cleaned with standard standard Environmental Protection Agency registered disinfectants.
- Group 2 Enhanced Standard: Trainees received the components of the Standard group and were instructed to take an additional 10-minute shower with soap and a wash cloth every week. They were also issued a first aid kit. Supplemental SSTI education for trainees and drill sergeants was also provided (e.g., pocket cards, posters). Drill sergeants received briefings on SSTI and skin inspection/minor wound care.
Period: Overall Study
Arm/Group | Group 1 Standard | Group 2 Enhanced Standard | Group 3 Chlorhexidine
Started | 9315 | 10864 | 10030
Completed | 8155 | 9250 | 8846
Not Completed | 1160 | 1614 | 1184
Not completed — Lost to Follow-up | 1160 | 1614 | 1184

BASELINE CHARACTERISTICS:
Population: Participants that developed SSTI.
Groups:
- Group 1 Standard: Trainees received a preventive medicine briefing augmented with SSTI and MRSA SSTI prevention information and personal hygiene instructions. Trainees seeking medical care for an SSTI received standardized SSTI care (e.g., antimicrobial therapy, wound management, patient education) at the Troop Medical Clinic. High-touch common surfaces within the battalion areas were cleaned with standard Environmental Protection Agency registered disinfectants.
- Total: Total of all reporting groups
Arm/Group | Group 1 Standard | Group 2 Enhanced Standard | Group 3 Chlorhexidine | Total
Number analyzed (Participants) | 303 | 439 | 461 | 1203
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.4 (3.1) | 20.3 (3.2) | 20.3 (2.9) | 20.3 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 303 | 439 | 461 | 1203
Race/Ethnicity, Customized [Number; unit: participants]
  White, non-Hispanic | 92 | 167 | 172 | 431
  Hispanic | 13 | 24 | 18 | 55
  Black, non-Hispanic | 7 | 7 | 4 | 18
  Other, non-Hispanic | 5 | 8 | 5 | 18
  Unknown | 186 | 233 | 262 | 681

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Skin and Soft Tissue Infection (SSTI)
Time Frame: At the end of the 20 month study
Measure: Number; unit: participants
Groups:
- Group 1 Standard: Trainees received a preventive medicine briefing augmented with SSTI and MRSA SSTI prevention information and personal hygiene instructions. Trainees seeking medical care for an SSTI received standardized SSTI care (e.g., antimicrobial therapy, wound management, patient education) at the Troop Medical Clinic (TMC). High-touch common surfaces within the battalion areas were cleaned with standard Environmental Protection Agency-registered disinfectants.
Arm/Group | Group 1 Standard | Group 2 Enhanced Standard | Group 3 Chlorhexidine
Number analyzed (Participants) | 9,315 | 10,864 | 10,030
participants | 303 | 439 | 461

2. Primary Outcome: Incidence of Methicillin-resistant Staphylococcus Aureus (MRSA)-Associated SSTI
Time Frame: At the end of the 20 month study
Measure: Number; unit: participants
Arm/Group | Group 1 Standard | Group 2 Enhanced Standard | Group 3 Chlorhexidine
Number analyzed (Participants) | 9,315 | 10,864 | 10,030
participants | 86 | 135 | 95

ADVERSE EVENTS:
Arm/Group | Group 1 Standard | Group 2 Enhanced Standard | Group 3 Chlorhexidine
Serious Adverse Events (participants affected / at risk) | 0/9315 | 0/10864 | 0/10030
Other Adverse Events (participants affected / at risk) | 0/9315 | 0/10864 | 4/10030
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 Standard (N=9315) | Group 2 Enhanced Standard (N=10864) | Group 3 Chlorhexidine (N=10030)
Dermatitis due to soap (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No